CLINICAL TRIAL: NCT03946124
Title: Prevention of Fall in Older Adults With Overactive Bladdar
Brief Title: Fall Prevention in Older Adults With OAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 822377
Record Dates: First submitted 2019-04-17; First posted 2019-05-10 (Actual); Results first posted 2019-12-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Intervention Model Description: prospective cohort design examining effects in adults aged 65 and older with OAB undergoing treatment with medication in a clinical setting. A follow up period of 8 weeks has been selected because this is the period of maximal drop in adherence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fesoterodine (Other): Subjects (irrespective of preference) will receive a 90-day supply of open label fesoterodine 4 mg per day. Medication will start 1 week after the baseline visit. After 2 weeks of treatment, dose may be increased to 8 mg over the telephone based on symptom report. This dosing regimen is direct alignment with clinical care. Change of prescription to another anti-cholinergic may occur during the study period, if determined necessary by the physician.
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine, the drug used in this study, is an appropriate medication for routine and standard care of overactive bladder.

SUMMARY:
Though OAB treatment may improve physical activity, there is a lack of easily administered instruments for measuring physical activity in older adults. Aim is to validate instruments to measure physical activity and preference for medication, and to determine the effect of preference for anti-cholinergic medication on adherence, physical activity, and falls risk. It's plan a prospective cohort study of adults aged 65 or older with OAB undergoing treatment with anti-cholinergic medication.

DETAILED DESCRIPTION:
Older adults with overactive bladder (OAB) have reduced physical activity and are at increased risk for falls. Though recent studies suggest that treatment of OAB may improve physical activity, there is a lack of easily administered instruments for measuring physical activity in older adults. Furthermore, physical activity outcomes in older adults with OAB are affected by treatment preference and potential neurocognitive dysfunction caused by anti-cholinergic medication. The aims of the present proposal are 1) to validate an instrument to measure physical activity 2) to validate an instrument to measure preference for medication and 3) to determine the effect of preference for anti-cholinergic medication on adherence, physical activity, and falls risk. Plan: a prospective cohort study of adults aged 65 or older with OAB undergoing treatment with anti-cholinergic medication. The primary outcome will be physical activity measured using a self-reported instrument and accelerometer at baseline and 8 weeks after treatment. Secondary outcomes will be fall risk defined by changes in neurocognitive testing, urinary symptoms, and medication adherence at 8 weeks after treatment. The findings of this study could provide a paradigm shift in the management of older adults with OAB and at increased risk for falls.

ELIGIBILITY:
Inclusion Criteria:

adults aged 65 or older, urinary urgency of quite a bit severity or more on the Overactive Bladder Questionnaire-Short Form (OABq-SF), eligible for pharmacologic therapy for overactive bladder

Exclusion Criteria:

predominant stress incontinence (on UDI-6), current/recent use (6 m) or contraindication to anti-cholinergic medication, severe voiding difficulties, men on 5-alpha reductase inhibitors, severe neurologic disease, recent anti-incontinence or prolapse surgery, other urinary tract conditions such as calculus or recurrent UTI.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Female
Enrollment: 74 (Actual)
Dates: Start 2015-07-25 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chu CM, Harvie H, Arya LA, Andy UU. Short-Term Effect of Fesoterodine on Physical Function Relevant to Fall Risk in Older Women With Overactive Bladder. Female Pelvic Med Reconstr Surg. 2021 Dec 1;27(12):759-765. doi: 10.1097/SPV.0000000000001046. PMID 34807883

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fesoterodine
Started | 74
Completed | 55
Not Completed | 19
Not completed — Withdrawal by Subject | 19

BASELINE CHARACTERISTICS:
Arm/Group | Fesoterodine
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 74
Physical Activity - Daily Steps [Median (Inter-Quartile Range); unit: Steps per day] | 2117.7 [988.5 to 2924.25]
Physical Activity - CHAMPS questionnaire caloric expenditure/week, all activities [Mean (Standard Deviation); unit: Kcal/week] | 2552.4 (2560.12)
Physical Activity - IPAQ questionnaire total physical activity [Mean (Standard Deviation); unit: MET-min/wk] | 785.62 (1609.84)
Short Physical Performance Battery total score [Mean (Standard Deviation); unit: units on a scale] — The short physical performance battery (SPPB) is a combination measure that examines gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and measures physical function in older people.
  Score 0-12. Higher scores mean better lower extremity function.
  units on a scale | 7.82 (2.21)
Mini Cog screening test [Count of Participants; unit: Participants] — The Mini Cog screening test consists of a 3-item recall test for memory and a clock drawing test. A score of <3 is considered a positive screen for cognitive impairment. Population: Not all patients completed baseline Mini Cog testing
  Participants
    number analyzed (Participants) | 68
    Normal cognition | 60
    Abnormal cognition | 8
OABq-SF Symptoms Severity score [Mean (Standard Deviation); unit: units on a scale] — The OABq-SF 19 item validated questionnaire that measures the impact of OAB symptoms on health-related quality of life and bother. Total scores range 0 to 100, with higher scores reflecting greater symptoms.
  units on a scale | 61.9 (23.8)
UDI-6 total score [Mean (Standard Deviation); unit: units on a scale] — The UDI-6 is a validated questionnaire that measures the impact of urinary incontinence on quality of life. Scores range from 0-100, with higher scores indicating higher bother from urinary incontinence.
  units on a scale | 44.2 (20.5)

OUTCOME MEASURES:

1. Primary Outcome: Measure of Physical Activity
Description: Physical activity was measured by using accelerometer worn over the course of a week at follow up. Average daily step counts were derived from this weeklong measurement.
Time Frame: 1 week
Population: Patients who were present at follow up and completed accelerometer wear were included in analysis.
Measure: Median (Inter-Quartile Range); unit: steps per day
Arm/Group | Fesoterodine
Number analyzed (Participants) | 56
steps per day | 1634.19 [980.1 to 2367.3]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Fesoterodine
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 7/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fesoterodine (N=74)
Side effects (Gastrointestinal disorders) | 6 (6) — Patients who experienced expected side effects of medication, including constipation, dry eyes, and dry mouth
Dizziness, edema (Vascular disorders) | 1 (1) — Patients who reported side effects not typically associated with fesoterodine, such as dizziness and edema. One subject experienced both AEs concurrently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT03946124/Prot_SAP_001.pdf
  • Informed Consent Form (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03946124/ICF_000.pdf